CLINICAL TRIAL: NCT01517646
Title: Pilot Study of CoolTXT for Non-Invasive Fat Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA11-003
Record Dates: First submitted 2012-01-04; First posted 2012-01-25 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2012-01

CONDITIONS: Body Fat Disorder
Keywords: Lipolysis; Cryolipolysis; Fat Reduction
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fat Reduction (No Intervention)
  Interventions: Device: The Zeltiq System

INTERVENTIONS:
Device: The Zeltiq System — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis; Lipolysis

SUMMARY:
This study is being performed to reduce unwanted fat, in various body areas, using a new applicator and control unit for Zeltiq.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and feasibility of a new product under development for non-invasive fat reduction. The new product delivers controlled cooling via a conformable surface applicator, rather than the existing vacuum applicator. A range of treatment parameters will be investigated. At the investigator's discretion, each treatment area may receive up to 3 treatments, spaced 2 - 8 weeks apart. The subjects will return for follow-up at 2 months and 4 months after final treatment. Therefore, the entire study period may last up to 8 months.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects > 18 years of age and < 65 years of age.
* Subject has clearly visible fat on intended treatment area(s), which in the investigator's opinion, may benefit from the treatment(s). Treatment areas include: abdomen, saddlebag (outer aspect of upper thighs), upper arms and inner thighs.
* Subject has not had weight change exceeding 10 pounds in the preceding month.
* Subject with body mass index (BMI) between 25 and 35. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
* Subject agrees to maintain his/her weight (i.e., within 5 pounds) by not making any major changes in their diet or lifestyle during the course of the study.
* Subject has read and signed a written informed consent form.

Exclusion Criteria

* Subject has had a surgical procedure(s) in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, abdominoplasty, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 6 months.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
* Subject is pregnant or intending to become pregnant in the next 8months.
* Subject is lactating or has been lactating in the past 6 months.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Efficacy Assessment through Ultrasound Measurements | 16 weeks post final treatment
  The primary endpoint will be analyzed by percent reduction in fat layer thickness, as measured by ultrasound.
  • Safety endpoint: incidence of device- or procedure-related adverse events. Acceptance criteria - zero incidences of UADEs.

SECONDARY OUTCOMES:
Outcome Measured by Photo Review and Subject Satisfaction Questionnaire | 16 weeks post final treatment
  * Comparison of pre- and 16-week post final treatment photographs of the treatment area(s).
  * Subject satisfaction as assessed by questionnaires administered at 16 weeks post final treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Boey, MD, Principal Investigator — Arbutus Laser Centre
Locations (1):
- Arbutus Laser Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No